CLINICAL TRIAL: NCT00874250
Title: An Evaluation of the GORE Conformable TAG® Thoracic Endoprosthesis for the Primary Treatment of Aneurysm of the Descending Thoracic Aortic
Brief Title: Thoracic Endoprosthesis for Treatment of Aneurysm of the Descending Thoracic Aortic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAG 08-03
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE CTAG Device (Experimental): The primary endpoint of this study is freedom from a Major Device Event (MDE) through 1 month post-treatment in subjects treated with the GORE® Conformable TAG® Thoracic Endoprosthesis.
  Interventions: Device: GORE CTAG Device

INTERVENTIONS:
Device: GORE CTAG Device — Endovascular aortic stent-graft
  Other Names: GORE Conformable TAG® Thoracic Endoprosthesis

SUMMARY:
To assess the safety and efficacy of the GORE Conformable TAG® Thoracic Endoprosthesis in the primary treatment of aneurysm of the descending thoracic aorta (DTA)

> Primary Hypothesis: The proportion of subjects free from a major device event through 1 month post-treatment will not be significantly less than 0.95, which represents the proportion observed in previous clinical studies with the GORE TAG® Thoracic Endoprosthesis

ELIGIBILITY:
Inclusion Criteria:>

1. Presence of DTA aneurysm deemed to warrant surgical repair >

* Fusiform (≥50 mm), or >
* Saccular (no diameter criteria)> 2. Subject is > 21 years of age> 3. Proximal and distal landing zone length ≥ 2.0 cm >
* Landing zones must be in native aorta>
* Landing zone may include left subclavian artery, if necessary> 4. All proximal and distal landing zone inner diameters are between 16-42 mm>
* Diameter assessed by flow lumen and thrombus, if present; calcium excluded> 5. Life expectancy > 2 years> 6. Able to tolerate thoracotomy > 7. Male or infertile female> 8. Able to comply with protocol requirements including following-up> 9. Signed informed consent>

Exclusion Criteria:>

1. Differing proximal and distal neck diameters (aortic taper) outside the intended aortic diameter requirements (sizing guide) for a single endoprosthesis diameter and the inability to use devices of different diameters (in adherence to the sizing guide) to compensate for the taper>
2. Tortuous or stenotic iliac and/or femoral arteries and inability to use a conduit for vascular access>
3. Aneurysmal, dissected, heavily calcified, or heavily thrombosed landing zone(s)>
4. Mycotic aneurysm>
5. Hemodynamically unstable aneurysm rupture>
6. Aortic dissection>
7. Planned coverage of left carotid or celiac arteries with the CTAG Device>
8. Planned concomitant surgical procedure (other than left subclavian transposition and wireless sac pressure monitoring), or major surgery within 30 days of treatment date>
9. Known degenerative connective tissue disease, e.g. Marfan or Ehler-Danlos Syndrome>
10. Known history of drug abuse>
11. ASA risk classification = V (moribund patient not expected to live 24 hours with or without operation)>
12. NYHA class IV >
13. Participating in another investigational device or drug study within 1 year of treatment>
14. Subject has known sensitivities or allergies to the device materials>
15. Subject has a systemic infection and may be at increased risk of endovascular graft infection>

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Jordan, Dr., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Medical Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordan WD, Desai N, Letter AJ, Matsumura JS. Long-term outcomes of the conformable TAG thoracic endoprosthesis in a prospective multicenter trial. J Vasc Surg. 2021 Nov;74(5):1491-1498. doi: 10.1016/j.jvs.2021.04.063. Epub 2021 May 20. PMID 34022380
- [Derived] Panthofer AM, Olson SL, Harris DG, Matsumura JS. Derivation and validation of thoracic sarcopenia assessment in patients undergoing thoracic endovascular aortic repair. J Vasc Surg. 2019 May;69(5):1379-1386. doi: 10.1016/j.jvs.2018.08.180. Epub 2018 Dec 28. PMID 30598352

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE CTAG Device
Started | 51
Completed | 0
Not Completed | 51

BASELINE CHARACTERISTICS:
Arm/Group | GORE CTAG Device
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Free From a Major Device Event Through 1 Month Post-treatment
Time Frame: Treatment through 1 month post treatment
Measure: Number; unit: participants
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
participants | 50 [50 to 50]
Statistical Analysis 1: Comparison: CTAG Device Aneurysym Subjects; Test type: Superiority or Other; p = 0.0024, Binomial Test; Proportion = 0.98, 95% CI 2-sided [0.895 to 0.996]

2. Secondary Outcome: The Number of Subjects Experiencing a Serious Adverse Event Through One Month Post Treatment.
Time Frame: Treatment through 1 month post procedure
Measure: Number; unit: participants
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
participants | 13

3. Secondary Outcome: Procedure Time (Minutes)
Description: Total time in minutes required for surgical device implantation.
Time Frame: Initial Device Implant Procedure During Index Hospitalization
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
Minutes | 118 [109.5 to 140.4]

4. Secondary Outcome: Operative Blood Loss (mL)
Description: Blood loss in mL during initial device implantation procedure
Time Frame: Initial Device Implant Procedure During Index Hospitalization
Measure: Median (Standard Deviation); unit: mL
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
mL | 150 (403.5)

5. Secondary Outcome: Days of Convalescence Stay in an Intensive Care Unit
Description: Convalescence stay (days) in an Intensive Care Unit during the initial hospitalization for the device implantation
Time Frame: During the Index Hospitalization
Measure: Number; unit: participants
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
participants | 38

6. Secondary Outcome: Total Length of Hospital Stay (Days)
Description: Total days of hospital stay during the initial hospitalization for implantation of device
Time Frame: Total Duration of the Index Hospitalization
Measure: Median (Full Range); unit: Days
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 51
Days | 4 [1 to 68]

7. Secondary Outcome: Time in Days to Return to Normal Daily Activities
Description: This is the self reported time (in days) that the subject returned to pre-operative activities and is not a time to event analysis.
Time Frame: Average time within one month window
Measure: Median (Full Range); unit: Days
Arm/Group | CTAG Device Aneurysym Subjects
Number analyzed (Participants) | 47
Days | 31 [3 to 374]

8. Secondary Outcome: Procedural Survival
Description: Subjects who survived the index procedure
Time Frame: Initial Device Implant Procedure During Index Hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | GORE CTAG Device
Number analyzed (Participants) | 51
Participants | 51

9. Secondary Outcome: Intensive Care Unit (ICU) Stay
Description: Subjects admitted to ICU during index hospitalization
Time Frame: Initial Device Implant Index Hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | GORE CTAG Device
Number analyzed (Participants) | 51
Participants | 38

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | CTAG Device Aneurysm Subjects
All-Cause Mortality (participants affected / at risk) | 19/51
Serious Adverse Events (participants affected / at risk) | 37/51
Other Adverse Events (participants affected / at risk) | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTAG Device Aneurysm Subjects (N=51)
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 5
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Neurogenic bowel (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Multimorbidity (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Stent-graft endoleak (General disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Gallbladder necrosis (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Sepsis (Infections and infestations) | 2
Sepsis syndrome (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Arterial injury (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
International normalised ratio increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Spinal cord disorder (Nervous system disorders) | 1
Spinal cord ischaemia (Nervous system disorders) | 1
Spinal epidural haematoma (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Accelerated hypertension (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 3
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic dissection rupture (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypoperfusion (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Iliac artery occlusion (Vascular disorders) | 2
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTAG Device Aneurysm Subjects (N=51)
Anaemia (Blood and lymphatic system disorders) | 18
Leukocytosis (Blood and lymphatic system disorders) | 3
Angina pectoris (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 8
Cardiac failure congestive (Cardiac disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 3
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 5
Stent-graft endoleak (General disorders) | 10
Bronchitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 4
Incision site pain (Injury, poisoning and procedural complications) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Mental status changes (Psychiatric disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10
Aortic aneurysm (Vascular disorders) | 3
Haematoma (Vascular disorders) | 5
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.